CLINICAL TRIAL: NCT06846788
Title: Can Physical Exercise Improve Sensory Outcome and Reduce Pain After Peripheral Nerve Injury in the Arm and Hand? - A Feasibility Study
Brief Title: Study of Nerve Injuries and Physical Exercise
Acronym: SNIPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Cecilia Mellstrand Navarro, ass professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-05306-01
Record Dates: First submitted 2025-01-17; First posted 2025-02-26 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Nerve Injury; Pain Management; Sensorial Disturbance
Keywords: physical exercise; sensory relearning; physical therapy; occupational therapy; hand surgery; nerve injury; pain management
MeSH Terms: conditions — Agnosia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical exercise (Experimental): The participants will perform supervised physical exercise on a stationary exercise bike, 30 minutes, 2 times a week, for 6 weeks. The exercise will be at moderate intensity (40-59 % VO2max).
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — A traditional sensory relearning rehab session will be performed after our intervention consisting of 30 minutes of physical exercise.
  Other Names: Aerob exercise; sensory relearning

SUMMARY:
This study will explore if combining exercise with sensory training can help improve sensory function and reduce pain after an injury to the nerves in the arm and hand. The study will look at how exercise affects the BDNF protein (which helps nerves grow), how it impacts sensation, and how it might help manage pain. Research has shown that exercise is good for brain health, enhancing abilities such as focus, memory, and the ability to cope with stress. It also helps the brain release BDNF, which helps nerve cell growth and plasticity. Higher levels of BDNF might improve sensory function, but no previous study has investigated the combination of exercise and sensory training.

Study aims to investigate:

* if it is possible to use a physical exercise program (using an exercise bike) for people with nerve injuries.
* how easy it is to recruit participants, how well they stick to the program
* if exercise can change BDNF levels and VO2max (a measure of fitness), and how these changes might relate to pain and sensory.
* if it's possible to run a bigger, more detailed study in the future and check if it could be helpful for patients.

The researchers believe that combining exercise with sensory training could help reduce pain and improve sensation compared to traditional sensory training methods.

Participants will:

* perform 30 minutes of exercise on a stationary bike, twice a week, for 6 weeks at a moderate level of effort. After the exercise, they will do 5-10 minutes of sensory training, with additional exercises to practice at home. The sensory training will follow a standard program designed to help retrain the brain to process sensory information.
* be subject to a blood sample Results will include sensory function, pain evaluation, patient reported outcome measures.

DETAILED DESCRIPTION:
Hypothesis The hypothesis posits that integrating physical exercise with sensory relearning may lead to a reduction in pain and an improvement in sensory interpretation. Potentially, adding physical activity both during the early and later stages of rehabilitation following PNI in the arm and hand could be beneficial, in comparison to only conventional sensory relearning. This study is planned as a feasibility study to investigate the possibility of using physical activity. The results, knowledge and insights from this study will be used in the design of a future RCT study at our clinic.

Aim The primary aim of this study is to evaluate the feasibility of implementing a structured physical activity program, using an exercise bike, after PNI in the arm and hand in a rehabilitation setting at the hand surgery department at Sodersjukhuset. The study is set out to assess the recruitment, retention rates and possible outcome measures, prior to design of a RCT. Further, the study will explore the responsiveness in pre- and post-intervention testing and the acceptability in the outcome measures. It will explore potential trends in BNDF and Vo2max changes and its potential correlation with pain and sensory function.

Study population

Recruitment of study population Patients with pain and/or decreased sensory function after a PNI in the arm and hand will be included. Health care practitioners at the department of Hand Surgery at Sodersjukhuset will identify potential participants that meet the study inclusion criteria either through search of medical journals or during visits at the hand surgery unit. An invitational letter with a description of study including a letter of consent will be handed to the patient personally or by mail and we will follow up with a telephone call. Intervention The participants will perform supervised physical exercise on a stationary exercise bike, 30 minutes, 2 times a week, for 6 weeks. The exercise will be at moderate intensity (40-59 % VO2max). The exercise will be held at the department of hand surgery at Sodersjukhuset, supervised by a physiotherapist. The intervention will be modified according to the physical ability of the participant. Immediately after the exercise, sensory relearning exercises will be performed for about 5-10 minutes. In addition, the participants will perform the sensory relearning at home. To conduct sensory relearning in brief periods at home, 4-5 times a day has been shown to be effective in previous studies following median nerve injuries (25). Multisensory early sensory relearning is carried out according to standardized sensory relearning protocol, appendix 1, (Kansletraningsinformation). Organization of the work The intervention starts with a familiarization session and introduction to the testing procedures and equipment. Oral and written information regarding the study will be provided by the treating therapist and a written consent will be obtained before the familiarization session starts. The questionnaires will be sent out before the first study visit. Baseline measures will be taken during session number two and will be conducted by the physiotherapist and co-researcher. The same procedure with measurements will be conducted after 6 weeks and a follow up at 12 weeks, see timeline (appendix 2 Flowchart). Baseline measures for BDNF will be measured before and after the first bike session at 3, 6, and 12 weeks. At each time point, a nurse will draw 10 mL blood sample and divide it into two separate containers (a heparinixed tube for plasma and a clot activator tube for serum analysis). The blood collected for plasma will be centrifuged at 6000 rpm (revolutions per minute) for 3 min, to separate the plasma while the tube for serum analysis will be left for at least 30 min to clot at room temperature, before being centrifuged at 6000 rpm for 15 min to separate the serum. Thereafter, both separated plasma and serum samples will be transferred to Eppendorf tubes, pseudonymized and provided with a code at the hand surgery department Södersjukhuset. The samples will then be transported to The Swedish School of Sport and Health Sciences where they will be stored at -80°C until analysis. Neurotrohic factors will be analysed using ELISA kits following the manufacturer´s instructions.

All the questionnaires will be sent out prior to the study by mail or electronically. All tests will be performed: Before intervention, 3 weeks, 6 weeks and 12 weeks.

Drop out and study adherence will be investigated with open-ended questions e.g. describe in your own words why you decided to end/continue the study participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral nerve in the arm and hand, treated at the rehabilitation unit at Södersjukhuset, between 2010-2025
* 14 days to 15 years after injury.
* Age above 18.

Exclusion Criteria:

* Psychiatric illness or substance addiction severe enough to make intervention impossible.
* Severe neurological disease.
* Severe diabetes mellitus with nerve complications.
* Severe cardiovascular disease where aerobic exercise is contraindicated.
* Unwillingness or medical inability to undergo the intervention.
* Insufficient knowledge of the Swedish or English language, which makes examination with patient-reported questionnaires impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility recruitment rate | 12 weeks
  Number of participants recruited per month.

SECONDARY OUTCOMES:
Change in interpretation of sensation in the hand measured with Static two-point discrimination (S2PD) using millimetres | first session, 3 weeks, 6 weeks and 12 weeks
  Static Two-Point Discrimination (S2PD) measures the minimum distance between two stimuli at which a patient can correctly identify them as distinct points. The recommendations of Moberg will be used where a light pressure of the instrument is exerted until blanching occurs. The prongs on the discriminator are applied longitudinally and perpendicular to the finger tips with one or two prongs, distance is measured in millimetres. 7 out of 10 correct answers are needed. The S2PD test will be used to describe one aspect of tactile gnosis, discriminative touch and to monitor if progression of functional sensibility is present. Individual change will be calculated in millimetres, as post cycle intervention millimetre -millimetre. S2PD will be measured before cycling intervention at 3, weeks 6 weeks and at follow up 12 weeks.
Evaluate potential recovery or regeneration of nerve function Semmes-Weinstein Monofilament (SWM) | first session, 3 weeks, 6 weeks and 12 weeks
  The Semmes-Weinstein monofilaments test (SWM) assess the threshold for perception of touch, which reflects re-innervation of cutaneous peripheral receptors. The test is used by applying nylon monofilaments of varying thickness to the skin to determine the minimum force required for detection. The test includes a set of monofilaments that correspond to different pressure thresholds, with thicker filaments indicating greater sensory impairment. SWM assess the threshold for perception of touch, which will be used to reflect re-innervation of cutaneous peripheral end organs. Measured in grams of pressure will be done to evaluate change. 5 pocket filaments from 70 miligrams to 300-450 grams will be used. The results from SWM are interpreted as being normal if the patient perceives ≤ 0.068 grams of pressure (filament number 2.83). Individual changes in sensory thresholds will be calculated by comparing pre-intervention SWM grams with those at 6 and 12 weeks.
Retention and adherence to intervention | At first session and continuously to 12 weeks
  The proportion of recruited participants able to cycle for 30 minutes without triggering pain and able and willing to continue the intervention calculated as the number of recruited participants able to cycle for 30 minutes without triggering pain and able and willing to continue the intervention divided by the total number of recruited participants.
Explore design and outcome measures | 12 weeks
  To investigate accessibility of outcome measures. Relevance to the participants will be asked and time in minutes it takes to fill out forms, sensory testing and the logistics of laboratory testing.
Explore trial design | 12 weeks
  Presented as the proportion of variables investigated and completed divided of the total number of variables.
Useful change in ability to identify objects with Shape Texture Identification (STI) | first session, 3 weeks, 6 weeks and 12 weeks
  The Shape/texture identification test (STI) consists of two subtests 1. Identification of three shapes; cube, cylinder or hexagon and 2. Identification of three textures; one, two or three raised metal dots placed in a row. The test includes three levels of difficulty by decreasing sizes of shapes and distance of dots. The score range from 0-6 with 0-3 on each subtest. A total score of 6 represent normal somatosensory function. The test is a sensory test for interpretation of tactile input. The test requires active manipulation and takes active touch into account. We aim to assess STI at baseline and to evaluate individual changes in somatosensory function after a 6-week cycling intervention (twice per week) and at a 12-week follow-up.
Change in neuropathic pain with Pain Douleur Neuropathique en 4 Questions (DN4) | Baseline, 3 weeks, 6 weeks, 12 weeks
  Neuropathic Pain Symptom Inventory DN4 will be used to identify neuropathic pain and to assess individual-level of changes in neuropathic pain symptoms. DN4 consists of 10 items (items 1-7 consists of self-report items about pain descriptors and 3 items are based on clinical examination. A score ≥4 suggests neuropathic pain. Individual change will be calculated as post-cycling intervention DN4 Score - Baseline DN4 Score, before cycling interventions measured at 6 weeks and at follow up 12 weeks will be evaluated individual. Negative values indicate improvement with a reduction in neuropathic symptoms.
Existing and changed anxiety and depressioin HADS (The Hospital Anxiety and Depression Scale) | first session, 3 weeks, 6 weeks and 12 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a self-assessment questionnaire with seven items for depression and seven for anxiety. Each item is scored from 0-3 (0 means 'no symptoms' and 3 'severe symptoms'). Scores range from 0-21 in each subscale. A high score indicates high level of anxiety or depression. A score ≥ 8 suggests that a disorder might exists, ≥ 11 suggests that depressive or anxiety disorder exists. We will measure individual change in HADS scores over three time points, calculate the total score for anxiety and depression at each assessment. Compare the scores over time to identify increases, decreases, or stability in symptoms. A meaningful change is typically considered a shift of ≥ 1.5 to 2 points in the subscale scores.
Patient questionnaire HQ8 (arm/hand) change over time | first session, 3 weeks, 6weeks and 12 weeks
  Patient questionnaire HQ8 (arm/hand) includes eight questions on perceived symptoms in the affected/operated hand (pain on load, pain on motion without load, pain at rest, stiffness, weakness, numbness, and cold sensitivity) and one question on the ability to perform activities of daily living. The questions are reported on a Likert scale (0-100) in ten-point increments. Zero represents no problem and 100 the worst problem imaginable
Pain VAS (The visual analog scale) | From the first bike session to the end of 12 weeks.
  the Visual Analog Scale (VAS) will be used before and during the cycling intervention to guide resistance levels and monitor any increase in pain in the arm/hand or other areas, thereby helping to limit adverse events.
Exertion rate during exercises, Borg Rating of Perceived Exertion (RPE) | From the first bike session to the end of 12 weeks.
  Borg Rating of Perceived Exertion (RPE) Scale allows individuals to rate their perceived level of exertion during the exercise. To guide the intervention. The scale is used to measure the intensity of exercise while on the bike, based on the physical sensations a person experiences, including increased heart rate, breathing rate, sweating, and muscle fatigue
Change in physical function and symptoms Quick DASH | Baseline, 3 weeks, 6 weeks and 12 weeks
  The Quick Disability of the Arm, Shoulder, and Hand (Quick DASH) is a self-reported instrument composed of eleven items. Six items measuring difficulties in physical activity due to upper extremity problems, two reflect severity of pain and tingling, three symptom items. The responses are rated on a 5-point Likert scale (1 = no difficulty, 5 = extreme difficulty). The total score ranges from 0-100, the higher score the more disability, regardless of which hand or arm the patient use. Individual changes in upper limb function using the Quick DASH questionnaire will be used at baseline, 3 weeks, after a 6-weeks of cycling intervention (twice per week) and at a 12-week follow-up.
Change in health-related quality of life | first session, 3 weeks, 6 weeks and 12 weeks
  The EQ-5D-5L measures health-related quality of life across five dimensions, each rated on a five-level severity scale. Responses are coded into a 5-digit health state, which requires a value set to generate a summary index score. Unlike simple summation, these numbers are labels without arithmetic properties. Additionally, the EQ VAS provides a self-rated health score from 0 to 100. The EQ-5D-5L will be used to quantify changes in an individual's health-related quality of life during the intervention by assessing five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) across five severity levels. This will be measured at baseline, 3 weeks, after a 6-week cycling intervention (twice per week) and at a 12-week follow-up.
  By comparing an individual's scores at different time points, improvements or deteriorations in health status can be identified and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia C Mellstrand Navarro, hand surgeon, ass professor, Principal Investigator — Department of Clinical Science and Education, Karolinska Institutet, Department of Hand Surgery, Södersjukhuset Hospital, and Department of Clinical Sciences Danderyd Hospital, Karolinska Institutet, Section for Orthopaedics, Stockholm, Sweden
Locations (1):
- Handkirurgiska kliniken Södersjukhuset, Stockholm, Sweden, Sweden

IPD SHARING:
Plan to Share IPD: No